CLINICAL TRIAL: NCT04439045
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study: Efficacy and Safety of VPM1002 in Reducing SARS-CoV-2 Infection Rate and COVID-19 Severity
Brief Title: Efficacy and Safety of VPM1002 in Reducing SARS-CoV-2 (COVID-19) Infection Rate and Severity
Acronym: COBRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Serum Institute of India Pvt. Ltd. (Industry); Max Planck Institute for Infection Biology (Other); Verity Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-5413
Record Dates: First submitted 2020-06-03; First posted 2020-06-19 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — VPM1002 recombinant BCG vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The clinical trial is designed as a double-blind (observer blind) study. Observer-blind means that during the course of trial, the companions/parents/guardians of the subjects and the study personnel responsible for the evaluation of any study endpoint will be unaware which vaccine was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VPM1002 (Experimental): A single dose of 0.1 mL of the reconstituted vaccine containing VPM1002 (Mycobacterium bovis rBCGΔureC::hly, live 2-8 × 105 CFU), administered via intradermal injection.
  Interventions: Biological: VPM1002
- Placebo (Placebo Comparator): A single dose of 0.1 mL of the 0.9% sodium chloride injection, administered via intradermal injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VPM1002 — VPM1002 is a recombinant BCG (rBCG)
  Other Names: Mycobacterium bovis rBCGΔureC::hly
  Arms: VPM1002
Other: Placebo — 0.9% sodium chloride
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
Bacille Calmette-Guerin (BCG) is a live attenuated vaccine administered for prevention of tuberculosis. Recently, several groups have hypothesized that BCG may "train" the immune system to respond to a variety of unrelated infections, including viruses and in particular the coronavirus responsible for COVID-19. Trials are currently being conducted in Australia, Netherlands, Germany and the United Kingdom to evaluate its effectiveness.

Front line workers includes members of municipal and provincial police services, emergency medical personnel, firefighters, public transport employees, health service workers and food manufacturing employees. They are at high risk of infection from COVID-19, with potentially high infection rate. The investigators propose an interventional trial to evaluate the effectiveness of BCG vaccination to prevent COVID-19 infection and reduce its severity in front-line employees in Ontario.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older
* Employee/member of: municipal or provincial police service, emergency medical services, fire services, public transport service, health service, food manufacturing facility

Exclusion Criteria:

* Prior intravesical BCG or intradermal BCG, with the exception of tuberculosis vaccination in childhood.
* Previous known history of latent or active tuberculosis
* Known kidney, liver or blood disorders which impairs organ and marrow function
* Chronic administration of steroids (>10 mg prednisone) at the time of randomization
* Current or planned concomitant biologic therapy in the next 7 months.
* Known hypersensitivity or allergy to components of VPM1002
* Pregnant or planning to become pregnant in the future 7 months.
* Breastfeeding.
* Current suspected viral or bacterial infection.
* Body temperature > 38° C
* Participation in another interventional study with potentially conflicting medication within 30 days before screening.
* The presence of an impaired immune response irrespective of whether this impairment is congenital or caused by disease, drugs or other therapy (e.g., anti-TNF therapy, methotrexate, azathioprine, antimalarials).
* Active malignancy requiring treatment.
* Known positive HIV serology.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BCG vaccine.
* Previous positive COVID-19 confirmed infection.
* Uncontrolled intercurrent illness.
* Psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
COVID-19 infection | 7 months
  To compare the self-reported incidence of SARS-CoV-2 infection (confirmed by positive test) following vaccination with either VPM1002 or placebo.

SECONDARY OUTCOMES:
Incidence of hospitalization for COVID-19 | 7 months
  To compare the incidence of hospitalization in participants with positive COVID-19 test treated with either VPM1002 or placebo
Incidence of ICU admission for COVID-19 | 7 months
  To compare the incidence of hospitalization requiring intensive care (ICU admission) in participants with positive COVID-19 test treated with either VPM1002 or placebo
Incidence of ARDS | 7 months
  To compare the incidence of acute respiratory distress syndrome (ARDS) in participants with positive COVID-19 test treated with either VPM1002 or placebo.
Mechanical ventilation for COVID-19 | 7 months
  To compare the incidence of the need for mechanical ventilation in participants with positive COVID-19 test treated with either VPM1002 or placebo.
Secondary infection in COVID-19 | 7 months
  To compare the incidence of secondary infection in participants with positive COVID-19 test treated with either VPM1002 or placebo.
COVID-19-related Mortality | 7 months
  To compare the mortality in participants with positive COVID-19 test treated with either VPM1002 or placebo.
Incidence of DVT | 7 months
  To compare the incidence of deep vein thrombosis, pulmonary embolism, or stroke in participants with positive COVID-19 test treated with either VPM1002 or placebo.

OTHER OUTCOMES:
Incidence of COVID-19 in Participants with Past BCG Vaccination | 7 months
  To compare the incidence of COVID-19 in participants who have received BCG vaccination previously vs those not previously vaccinated
Measure cardiac troponin, B-type natriuretic peptide, N-terminal pro b-type natriuretic peptide, C reactive protein, serum amyloid A, and procalcitonin as biomarkers of COVID-19 | 7 months
  To measure cardiac troponin, B-type natriuretic peptide, N-terminal pro b-type natriuretic peptide, C reactive protein, serum amyloid A, and procalcitonin identified as potential biomarkers of COVID-19 infection using blood samples collected prior to the vaccination and at the end of the 7-month follow-up.
Adverse events following BCG vaccine | 7 months
  To compare adverse event profile in participants following administration of VPM1002 or placebo when used for prevention of COVID-19.
Innate Trained Immunity | 7 months
  Compare the priming of the innate trained immunity (i.e. induction of Th1 and Th17 responses to unrelated stimuli) in participants following administration of VPM1002 or placebo when used for prevention of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre R Zlotta, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249